CLINICAL TRIAL: NCT02408718
Title: Assistive Device Training for Functional Mobility and Connectivity in Multiple Sclerosis
Brief Title: Assistive Device Training in Multiple Sclerosis
Acronym: ADT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Portland VA Medical Center (U.S. Federal Agency)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Michelle H. Cameron, MD, PT, MCR, Neurologist, Portland VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 3559
Record Dates: First submitted 2015-03-27; First posted 2015-04-03 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-04

CONDITIONS: Multiple Sclerosis
Keywords: Mobility; walking aids; falls; gait and balance
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Training group (Active Comparator): Subjects randomized to this group will receive a 6 week Assistive Device Training program in the use of their assistive device. They will have mobility assessments taken at baseline, after the training program has been completed, and 3 months later. During this time, their falls will be recorded monthly using prospective falls calendars. Members of this group will also receive MRI scans at baseline and after the completion of the training program.
  Interventions: Behavioral: Assistive Device Training
- Wait-list control (No Intervention): Subjects in this group will participate in the same mobility assessments and completion of the falls calendars, but will receive no intervention during this time. These subjects will have the opportunity to receive the training sessions when all assessment visits have been completed. These subjects will not receive MRI scans.

INTERVENTIONS:
Behavioral: Assistive Device Training — Six-week training program on the proper use of the subject's assistive device (eg. cane, walker, etc).
  Arms: Training group

SUMMARY:
The purpose of this study is to determine whether a training program in the use of ambulatory assistive devices (such as canes, walkers, etc) can reduce falls and increase functional mobility and neural connectivity in people with Multiple Sclerosis.

DETAILED DESCRIPTION:
40 people with Multiple Sclerosis, who routinely use ambulatory assistive devices and have fallen at least once in the past year, will be randomized into two groups. One group will receive a 6-week training program in the use of their assistive device; the other group will be wait-listed, and may choose to receive the training after their participation in the study is completed. All participants will receive mobility assessments at baseline, 6-8 weeks later, and 3 months after that. All participants will record their falls on falls calendars. Participants in the training group will receive MRI scans to assess neural connectivity at baseline and after completion of the training program.

The purpose of the study is to determine whether participation in the training program reduces falls and increases functional mobility when compared to the wait-listed group, and also to determine whether any change in neural connectivity, as assessed by MRI scans, is seen in those who participate in the training.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Sclerosis of any type,
* self-reported history of at least 1 fall in the previous year,
* able to walk at least 25 feet with or without an assistive device,
* clinically stable Multiple Sclerosis (no relapse in 30 days prior to enrollment),
* intermittent or constant unilateral or bilateral assistance required to walk,
* right-handed, willingness to remain consistent with medication use and level of physical activity for the duration of the study.

Exclusion Criteria:

* serious psychiatric or medical conditions that would preclude reliable participation in the study,
* dementia (MMSE <24),
* deafness,
* blindness,
* inability to follow directions in English,
* significant upper extremity tremor or weakness,
* more than 1 hour of assistive device training within the previous 3 years,
* any exclusions to receiving MRI scans (implanted devices, anxiety, claustrophobia, body weight over 350 lbs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Functional Mobility at Completion of Training and the Following Three Months | At baseline, 1 week after completion of training, 3 months later
  Timed Up and Go test, Timed 25-Foot Walk, 2 minute timed walk), Multiple Sclerosis Walking Scale-12
Change from Baseline in Falls at Completion of Training and the Following Three Months | First week of training, last week of training, 3 months later
  Change in rate of falls between time frames
Change from Baseline in Functional Neural Connectivity (fMRI) at Completion of Training | At baseline, 1 week after completion of training
  Resting-state (task free) functional Magnetic Resonance Imaging (fcMRI)

SECONDARY OUTCOMES:
Change from Baseline in Satisfaction with Assistive Device at Completion of Training and the Following Three Months | At baseline, 1 week after completion of training, 3 months later
  Quebec User Evaluation of Satisfaction with Assistive Technologies
Change from Baseline in Balance Confidence at Completion of Training and the Following Three Months | At baseline, 1 week after completion of training, 3 months later
  Activities-specific Balance Confidence Questionnaire
Change from Baseline in Multiple Sclerosis Impact at Completion of Training and the Following Three Months | At baseline, 1 week after completion of training, 3 months later
  Multiple Sclerosis Impact Scale-29
Change from Baseline in Physical Activity at Completion of Training and the Following Three Months | At baseline, 1 week after completion of training, 3 months later
  International Physical Activity Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Michelle H. Cameron, MD, PT MCR, Principal Investigator — Portland VA Medical Center
Locations (1):
- VA Portland Health Care System, Portland, Oregon, United States

REFERENCES:
- [Derived] Martini DN, Zeeboer E, Hildebrand A, Fling BW, Hugos CL, Cameron MH. ADSTEP: Preliminary Investigation of a Multicomponent Walking Aid Program in People With Multiple Sclerosis. Arch Phys Med Rehabil. 2018 Oct;99(10):2050-2058. doi: 10.1016/j.apmr.2018.05.023. Epub 2018 Jun 26. PMID 29958906